CLINICAL TRIAL: NCT06160232
Title: Psilocybin-Assisted Therapy for Severe Alcohol Use Disorder: Feasibility, Clinical Efficacy & (Neuro)Cognitive Mechanisms
Brief Title: Psilocybin-Assisted Therapy for Severe Alcohol Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Prof. Charles Kornreich, Head of Department of Psychiatry, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUB-Psy-PATh for sAUD; 2022-002369-14 (EudraCT Number)
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Severe Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized, double-blind, placebo-controlled, 1:1 parallel-group 7-month clinical trial comparing the effects of a high dose of psilocybin to those of a low dose of psilocybin (active placebo) provided within the context of a brief standardized psychotherapeutic intervention in 62 participants with severe alcohol use disorder.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high dose psilocybin (Experimental): 31 participants will receive a single administration of 30mg psilocybin provided within the context of a brief standardized psychotherapeutic intervention.
  Interventions: Drug: Psilocybin (high dose)
- low dose psilocybin (active placebo) (Placebo Comparator): 31 participants will receive a single administration of a very low dose of psilocybin (active placebo) provided within the context of a brief standardized psychotherapeutic intervention.
  Interventions: Drug: Active placebo (low dose of psilocybin)

INTERVENTIONS:
Drug: Psilocybin (high dose) — Psilocybin-assisted therapy
  Arms: high dose psilocybin
Drug: Active placebo (low dose of psilocybin) — Placebo-assisted therapy
  Arms: low dose psilocybin (active placebo)

SUMMARY:
Psilocybin-Assisted Therapy for Severe Alcohol Use Disorder: Protocol for a Double-Blind, Randomized, Placebo-Controlled, 7-month Parallel-Group Phase II Superiority Trial

DETAILED DESCRIPTION:
A substantial proportion of patients with alcohol use disorder does not respond to available treatments, which calls for the development of new alternatives. In parallel, psilocybin-assisted therapy for alcohol use disorder has recently yielded promising preliminary results. Building on extant findings, the proposed study aims to determine the feasibility and preliminary clinical efficacy of psilocybin-assisted therapy as a complementary intervention during inpatient rehabilitation for severe alcohol use disorder, and to characterize associated changes in the two key neurocognitive systems identified by dual-process models of addiction.

In this double-blind, randomized, placebo-controlled, 7-month parallel-group phase II superiority trial, 62 participants aged 21-64 years will be enrolled to undergo psilocybin-assisted therapy within the context of a 4-week inpatient rehabilitation for severe alcohol use disorder. The experimental group will receive a high dose of psilocybin (30 mg), whereas the control group will receive an active placebo dose of psilocybin, both within the context of a brief standardized psychotherapeutic intervention. The primary clinical outcome is the between-group difference in terms of the change in percentage of heavy drinking days from baseline to four weeks post-hospital discharge, whilst safety and feasibility metrics will also be reported as primary outcomes. Key secondary assessments include between-group differences in terms of changes in 1) drinking behavior parameters up to six months post-hospital discharge, 2) phosphatidyl-ethanol blood concentration, an objective biomarker of alcohol consumption, 3) symptoms of depression, anxiety, trauma, and global functioning, 4) neuroplasticity and key neurocognitive mechanisms associated with addiction, 5) psychological processes and alcohol-related parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 21 and 64 years old, with a BMI between 17.5 and 30 kg/m2 who
* Want to stop or decrease their drinking;
* Agree to have all psilocybin-assisted therapy sessions (preparation, administration, integration) and semi-structured interviews recorded;
* Have a diagnosis of Severe Alcohol Use Disorder (sAUD), according to the DSM-V (6 criteria or more), ascertained using the Mini International Neuropsychiatric Interview (M.I.N.I 7.0.2).
* Are not currently receiving any pharmacological treatment for sAUD and are willing to engage in all study requirements (including attending all study visits, preparatory sessions, integration sessions, follow-up sessions, and completing all study evaluations).
* Women of childbearing potential must have a negative serum pregnancy test at admission (day 1 +/-2) and a negative urine pregnancy test the day before psilocybin administration (day 19 +/-2).
* Women of childbearing potential must be using an effective, established method of contraception from inclusion until four weeks post-hospital discharge (5 weeks post-psilocybin administration). The following methods of contraception, if used properly and used for the duration of the study, are considered reliable: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: - oral, - intravaginal, - transdermal; progestogen-only hormonal contraception associated with inhibition of ovulation: - oral, - injectable, - implantable; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner (provided that partner is the sole sexual partner of the woman of child-bearing potential trial participant and that the vasectomised partner has received medical assessment of the surgical success; sexual abstinence (only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject). Note: female participants who are permanently sterilized (eg hysterectomy and/or bilateral salpingectomy) or post-menopausal (at least 48 consecutive weeks without menstruation) are not considered as being of child bearing potential.
* Men with a woman of childbearing potential partner should use a condom from inclusion until four weeks post-hospital discharge (5 weeks post-psilocybin administration).
* Good physical health with no unstable medical conditions, as determined by medical history, physical examination, routine blood labs, electrocardiogram, urine analysis, and urine toxicology.
* Willing to refrain from consuming psychoactive substances after enrolling in the study and during follow-up.
* Ability to provide voluntary written informed consent after receiving written information about the study protocol.
* Undergoing a 4-week alcohol detoxification program at the Brugmann University Hospital.
* Remaining abstinent from alcohol during the detoxification program (abstinence will be monitored using a breathalyzer during unannounced checks).
* Normal level of language comprehension (French).
* Affiliation to the Belgian social security system.

Exclusion Criteria:

* Allergy, hypersensitivity, or other adverse reactions to previous use of psilocybin or other hallucinogens.
* Uncorrected hypertension.
* Cardiovascular diseases, hepatic diseases, gastroenterological diseases, hematologic diseases, renal diseases, endocrine diseases, metabolic diseases, inflammatory diseases, neurological diseases or any other somatic condition that, in the opinion of the medical investigator (necessarily an M.D.), would pose a risk to the participant's participation in the study.
* Other somatic conditions that, in the opinion of the investigator, would pose a risk to the participant's participation in the study.
* Decompensated hepatic cirrhosis, defined by Child B or C score.
* Serious abnormalities of complete blood count or chemistries, biological abnormalities including TP < 50%, albumin < 35 g/L, total bilirubin > 35 μmol/L, leading to a Child B or C score.
* Abnormal ECG. Clinical ECG diagnoses and ECG signs subject to exclusion and needing medical attention: Atrial flutter or fibrillation, AV block 2nd degree or higher, AVNRT (AV-nodal re-entry tachycardia), AVRT (atrioventricular re-entry tachycardia), tri-fascicular block, signs of rare conditions such as Brugada syndrome or Wolff-Parkinson White Syndrome (Delta wave), Epsilon wave, Fusion beats, signs of acute myocardial ischemia such as ST elevation, signs of pulmonary embolism, Long QTc (≥470 ms for males and ≥480 ms for females), Sinus bradycardia <40bpm, Sinus node dysfunction (Sick sinus syndrome), Sinus node exit block, Supraventricular tachycardia (SVT), Torsades de Pointes, Ventricular fibrillation, Ventricular flutter, Ventricular tachycardia. This list might not be exhaustive and any other anomaly will be thoroughly assessed by the study physician, lead to exclusion if deemed necessary and referred to cardiology if warranted.
* Cognitive impairment (Folstein Mini Mental State Exam (Folstein et al., 1975) score < 26).
* Alcohol withdrawal complication(s), seizure, head injury or stroke within the last 6 months.
* Current active acute stress disorder/post-traumatic stress disorder,
* Lifetime history of schizophrenia spectrum disorders (schizophrenia, schizoaffective disorder, unspecified), other psychotic disorders or bipolar spectrum disorders (Type I, II, unspecified).
* Lifetime history of major depressive episode with psychotic features.
* Significant risk of suicide according to clinician assessment.
* Family history of schizophrenia spectrum disorders (schizophrenia, schizoaffective disorder, unspecified), or other psychotic disorders, or bipolar Type I in first- or second-degree relatives.
* Other substance use disorder (except for caffeine, nicotine, or cannabis) according to DSM-V criteria in the two months preceding inclusion to the study.
* Severe cannabis use disorder according to the DSM-V.
* Need to take medication with significant potential to interact with classical psychedelics (e.g., antidepressants except selective serotonin reuptake inhibitors (SSRIs), antipsychotics, psychostimulants, treatments for alcohol addiction as naltrexone or acamprosate or baclofen, opioid agonist treatment as buprenorphine or methadone, lithium, anticonvulsants, other dopaminergic or serotonergic agents, inhibitors of UGT1A9 and 1A10, monoamine oxidase inhibitors (MAOIs), aldehyde dehydrogenase inhibitors (ALDHs) and alcohol dehydrogenase inhibitors (ADHs)).
* High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, antisocial behavior, serious current stressors, lack of meaningful social support).
* History of hallucinogen use disorder, or >25 lifetime uses.
* Pregnancy and breastfeeding, at screening visit and till dosing day.
* Known or suspected non-compliance.
* Previous enrollment into the current study.
* Enrollment of the investigator, his/her family members, employees and other dependent persons.
* Patient subject to a legal protection measure (guardianship, curatorship or safeguard of justice), patient unable to express consent and not subject to a protection measure.
* Patients with language barrier (unable to follow the protocol or respond to clinical assessments).

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Primary clinical outcome: change in percentage of heavy drinking days | Baseline (going back to 8 weeks pre-enrolment) to 4 weeks post-hospital discharge
  The primary clinical outcome is the difference between the two treatment arms in terms of change from baseline (going back 8 weeks pre-enrolment) to 4 weeks post-hospital discharge (week 1 to 4 post-discharge) in the percentage of heavy drinking days. A heavy drinking day is defined as a day with ≥ 5 standard drinks/60g of alcohol for males, and ≥ 4 standard drinks/48g of alcohol for females. Alcohol consumption will be measured using the Timeline Follow-Back method (Sobell & Sobell, 1992), a semi-structured interview that provides estimates of the daily quantity, frequency, and pattern of alcohol (and other drugs) use during a set time period. The method has demonstrated adequate to excellent reliability and validity over a wide range of studies and clinical contexts (Carey, 1997; Sobell et al., 1996).
Feasibility: recruitment and retention rate | Recruitment rate: at screening and enrolment. Retention rate: at each study visit
  Recruitment and retention rate will be recorded and reported. A consort diagram displaying participant retention at each phase of the recruitment, screening and data collection process will be presented. We will report the numbers of individuals provided with participant information sheets who subsequently decided not to participate in the trial, number that underwent screening and number of drop-outs. For full transparency on inclusivity, information on the demographics and reason for exclusion will be reported from the screening dataset.
Safety: adverse events | At each study visit
  Adverse events will be systematically assessed at each study visit and follow-ups. Adverse events summary tables will display the total number of participants reporting an adverse event and the percentage of participants (%) with an adverse event.

SECONDARY OUTCOMES:
Percent Heavy Drinking Days | from pre-hospitalisation (up to 8 weeks pre-hospitalization) to 6 months post-hospital discharge (week 5 to 26 weeks)
  Alcohol consumption as measured with the Timeline Follow Back Method
Drinks per Day | from pre-hospitalisation (up to 8 weeks pre-hospitalization) to 4 weeks and 6 months post-hospital discharge
  Alcohol consumption as measured with the Timeline Follow Back Method
Percent Days Abstinent | from pre-hospitalisation (up to 8 weeks pre-hospitalization) to 4 weeks and 6 months post-hospital discharge
  Alcohol consumption as measured with the Timeline Follow Back Method
EEG-derived auditory long-term potentiation | Neuroplasticity EEG data will be collected pre-dosing and twice post-dosing (+1 day, +7 days)
  Index of cortical neuroplasticity
EEG-derived alcohol cue reactivity | EEG data will be collected pre-dosing and twice post-dosing (+1 day, +7 days)
EEG-derived inhibitory control | EEG data will be collected pre-dosing and twice post-dosing (+1 day, +7 days)
Psychological flexibility | Baseline, one day prior to psilocybin administration, one week post-psilocybin administration, as well as four weeks, three and six months post-hospital discharge.
  The Acceptance and Action Questionnaire II (AAQII; Bond et al., 2011)
Connectedness | Baseline, one day prior to psilocybin administration, one week post-psilocybin administration, as well as four weeks, three and six months post-hospital discharge.
  The Watts Connectedness Scale (WCS; Watts et al., 2022)
Interoception | Baseline, one day prior to psilocybin administration, one week post-psilocybin administration, as well as four weeks, three and six months post-hospital discharge.
  The Multidimensional Assessment of Interoceptive Awareness (MAIA; Mehling et al., 2012)
Depressive symptoms | Baseline, one day prior to psilocybin administration, one week post-psilocybin administration, as well as four weeks, three and six months post-hospital discharge.
  Beck Depression Inventory (BDI; Beck et al., 1961)
Anxiety symptoms | Baseline, one day prior to psilocybin administration, one week post-psilocybin administration, as well as four weeks, three and six months post-hospital discharge.
  StateTrait Anxiety Inventory - trait subscale (STAI; Spielberger et al., 1983)
Trauma symptoms | Baseline, one day prior to psilocybin administration, one week post-psilocybin administration, as well as four weeks, three and six months post-hospital discharge.
  International Trauma Questionnaire (ITQ; Cloitre et al., 2018)
Substance use recovery (patient reported outcome measure - PROM) | Baseline as well as four weeks, three and six months post-hospital discharge.
  Substance Use Recovery Evaluator (SURE; Neale et al., 2016)
Alcohol craving | Baseline, one day prior to psilocybin administration, one week post-psilocybin administration, as well as four weeks, three and six months post-hospital discharge.
  Penn Alcohol Craving Scale (PACS; Flannery et al., 1999)
Abstinence self-efficacy | Baseline, one day prior to psilocybin administration, one week post-psilocybin administration, as well as four weeks, three and six months post-hospital discharge.
  Alcohol Abstinence Self-Efficacy Scale (AASE; DiClemente et al., 1994)
Readiness to change | Baseline, one day prior to psilocybin administration, one week post-psilocybin administration, as well as four weeks, three and six months post-hospital discharge.
  Likert-scale ratings of the participant's perception of 1) the importance of change in drinking; 2) confidence of ability to change; 3) readiness for change; 4) Commitment to the goal of abstinence (Bogenschutz et al., 2022)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kornreich, M.D. Ph.D., Principal Investigator — Brugmann University Hospital, Free University of Brussels
Locations (1):
- Brugmann University Hospital, Brussels, Belgium

REFERENCES:
- [Background] Bogenschutz MP, Ross S, Bhatt S, Baron T, Forcehimes AA, Laska E, Mennenga SE, O'Donnell K, Owens LT, Podrebarac S, Rotrosen J, Tonigan JS, Worth L. Percentage of Heavy Drinking Days Following Psilocybin-Assisted Psychotherapy vs Placebo in the Treatment of Adult Patients With Alcohol Use Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Oct 1;79(10):953-962. doi: 10.1001/jamapsychiatry.2022.2096. PMID 36001306
- [Derived] Vanderijst L, Hever F, Buot A, Daure C, Benoit J, Hanak C, Veeser J, Morgieve M, Campanella S, Kornreich C, Mallet L, Leys C, Noel X. Psilocybin-assisted therapy for severe alcohol use disorder: protocol for a double-blind, randomized, placebo-controlled, 7-month parallel-group phase II superiority trial. BMC Psychiatry. 2024 Jan 26;24(1):77. doi: 10.1186/s12888-024-05502-y. PMID 38279085